CLINICAL TRIAL: NCT02127125
Title: Mechanism of Microbiome-induced Insulin Resistance in Humans (Aim2)
Acronym: MicroB2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC20130458H
Record Dates: First submitted 2014-04-24; First posted 2014-04-30 (Estimated); Results first posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-08

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — maltodextrin; Synbiotics; Sevelamer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Type2 Diabetes Mellitus - Placebo (Placebo Comparator): Type 2 Diabetes Mellitus subjects will receive maltodextrin (placebo)
  Interventions: Drug: Maltodextrin
- Obese with NGT - Placebo (Placebo Comparator): Obese (BMI = 30-37 kg/m2) normal glucose tolerant (NGT) subjects will receive maltodextrin (placebo)
  Interventions: Drug: Maltodextrin
- Lean with NGT -Placebo (Placebo Comparator): Lean (BMI< 26 kg/m2) normal glucose tolerant (NGT) will receive maltodextrin (placebo)
  Interventions: Drug: Maltodextrin
- Type2 Diabetes Mellitus - Synbiotic (Active Comparator): Type 2 Diabetic subjects will receive synbiotic
  Interventions: Drug: Synbiotic
- Type2 Diabetes Mellitus - Sevelamer (Active Comparator): Type 2 Diabetic subjects will receive sevelamer
  Interventions: Drug: Sevelamer
- Obese with NGT - Synbiotic (Active Comparator): Obese (BMI = 30-37 kg/m2) normal glucose tolerant subjects (NGT) will receive Synbiotic
  Interventions: Drug: Synbiotic
- Obese with NGT - Sevelamer (Active Comparator): Obese subjects (BMI = 30-37 kg/m2) normal glucose tolerant (NGT) will receive Sevelamer
  Interventions: Drug: Sevelamer
- Lean with NGT - Synbiotic (Active Comparator): Lean (BMI< 26 kg/m2) normal glucose tolerant (NGT) will receive Synbiotic
  Interventions: Drug: Synbiotic
- Lean with NGT - Sevelamer (Active Comparator): Lean (BMI< 26 kg/m2) normal glucose tolerant (NGT) will receive Sevelamer
  Interventions: Drug: Sevelamer

INTERVENTIONS:
Drug: Maltodextrin — Maltodextrin treatment as a placebo group. Maltodextrin, 6 gm three times a day for 4 weeks.
  Arms: Lean with NGT -Placebo; Obese with NGT - Placebo; Type2 Diabetes Mellitus - Placebo
Drug: Synbiotic — Synbiotic [5 g of oligofructose + 1 g Bifidobacterium longum R0175 (4 billion colony forming unit (CFU)/g) three times a day) for 4 weeks.
  Arms: Lean with NGT - Synbiotic; Obese with NGT - Synbiotic; Type2 Diabetes Mellitus - Synbiotic
Drug: Sevelamer — Sevelamer (1.6 g sevelamer + 4.4 g maltodextrin three times a day), for 4 weeks
  Other Names: Renvela
  Arms: Lean with NGT - Sevelamer; Obese with NGT - Sevelamer; Type2 Diabetes Mellitus - Sevelamer

SUMMARY:
The purpose of this study is to determine whether microbiome modulation and an experimental reduction in plasma LPS concentration improve inflammation and insulin action in insulin resistant (obese and T2DM) subjects.

DETAILED DESCRIPTION:
In this Aim we will test the hypothesis that lowering lipopolysaccharide (LPS) concentration in the circulation will improve systemic (muscle) inflammation and glucose metabolism in insulin resistant (obese and T2DM) subjects by protecting the intestinal barrier with a synbiotic (Bifidobacterium longum R0175 and oligofructose) or by sequestering LPS in the gastrointestinal lumen with sevelamer.

ELIGIBILITY:
Inclusion Criteria:

* Both genders (50%, male). All races and ethnic groups.
* Premenopausal women in the follicular phase, non-lactating, and with a negative pregnancy test. Postmenopausal women on stable dose of or not exposed to hormone replacement for ≥6 months.
* Hematocrit (HCT)≥ 34%, serum creatinine ≤ 1.4 mg/dl, and normal results of serum electrolytes, urinalysis, and coagulation tests. Liver function tests (LFTs) up to 2 times normal
* Stable body weight (±2%) for ≥ 3 months.
* Two or less sessions of strenuous exercise/wk for last 6 months.

Exclusion Criteria:

* Current treatment with drugs known to affect glucose and lipid homeostasis. If the subject has been on a stable dose for the past 3 months, the following agents will be permitted: calcium channel blockers, β-blockers, ACE inhibitors, angiotensin receptor blockers, and statins
* History of allergy to sevelamer.
* Non-steroidal anti-inflammatory drugs or systemic steroid use for more than a week within 3 months.
* Current treatment with anticoagulants (warfarin). Aspirin (up to 325 mg) and clopidogrel will be permitted if these can be held for seven days prior to the biopsy in accordance with the primary physician.
* Use of agents that affect gut flora (e.g. antibiotics, colestyramine, lactulose, PEG) within 3 months.
* History of heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the ECG), peripheral vascular disease, pulmonary disease, smokers.
* Poorly controlled blood pressure (systolic BP>170, diastolic BP>95 mmHg).
* Active inflammatory, autoimmune, hepatic, gastrointestinal, malignant, and psychiatric disease.
* History of gastrointestinal surgery or gastrointestinal obstruction within two years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Musi, MD., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Audie L. Murphy VA Hospital, STVHCS, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 69 participants were screened, 8 were screen failures, so not randomized.
Groups:
- Lean With NGT-Placebo: Lean (BMI< 26 kg/m2) normal glucose tolerant Maltodextrin treatment as a placebo group. Maltodextrin, 6 gm three times a day for 4 weeks.
- Lean With NGT-Sevelamer: Lean (BMI< 26 kg/m2) normal glucose tolerant Sevelamer (1.6 g sevelamer + 4.4 g maltodextrin three times a day), for 4 weeks
- Lean With NGT-Synbiotic: Lean (BMI< 26 kg/m2) normal glucose tolerant Synbiotic [5 g of oligofructose + 1 g Bifidobacterium longum R0175 (4 billion colony forming unit (CFU)/g) three times a day) for 4 weeks.
- Obese With NGT-Placebo: Obese (BMI = 30-37 kg/m2) normal glucose tolerant. Maltodextrin treatment as a placebo group. Maltodextrin, 6 gm three times a day for 4 weeks
- Obese With NGT-Sevelamer: Obese (BMI = 30-37 kg/m2) normal glucose tolerant. Sevelamer (1.6 g sevelamer + 4.4 g maltodextrin three times a day), for 4 weeks
- Obese With NGT-Synbiotic: Obese (BMI = 30-37 kg/m2) normal glucose tolerant. Synbiotic [5 g of oligofructose + 1 g Bifidobacterium longum R0175 (4 billion colony forming unit (CFU)/g) three times a day) for 4 weeks.
- Type 2 Diabetes -Placebo: Type 2 Diabetics Maltodextrin treatment as a placebo group. Maltodextrin, 6 gm three times a day for 4 weeks.
- Type 2 Diabetes-Sevelamer: Type 2 Diabetics Sevelamer (1.6 g sevelamer + 4.4 g maltodextrin three times a day), for 4 weeks
- Type 2 Diabetes-Synbiotic: Type 2 Diabetics Synbiotic [5 g of oligofructose + 1 g Bifidobacterium longum R0175 (4 billion colony forming unit (CFU)/g) three times a day) for 4 weeks.
Period: Overall Study
Arm/Group | Lean With NGT-Placebo | Lean With NGT-Sevelamer | Lean With NGT-Synbiotic | Obese With NGT-Placebo | Obese With NGT-Sevelamer | Obese With NGT-Synbiotic | Type 2 Diabetes -Placebo | Type 2 Diabetes-Sevelamer | Type 2 Diabetes-Synbiotic
Started (Passed screening for inclusion in study, assigned to intervention after baseline measurements.) | 6 | 8 | 9 | 11 | 12 | 12 | 2 | 0 | 1
Completed | 6 | 8 | 8 | 10 | 9 | 9 | 2 | 0 | 1
Not Completed | 0 | 0 | 1 | 1 | 3 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Low enrollment of Type 2 Diabetics in this study due to exclusionary medication criteria including many common diabetes medications such as metformin which interfere with microbiome content. Subjects were randomized to treatment and no diabetic subjects ended up in the sevelamer treatment group.
Groups:
- Type 2 Diabetes-Placebo: Type 2 Diabetics Maltodextrin treatment as a placebo group. Maltodextrin, 6 gm three times a day for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Lean With NGT-Placebo | Lean With NGT-Sevelamer | Lean With NGT-Synbiotic | Obese With NGT-Placebo | Obese With NGT-Sevelamer | Obese With NGT-Synbiotic | Type 2 Diabetes-Placebo | Type 2 Diabetes-Sevelamer | Type 2 Diabetes-Synbiotic | Total
Number analyzed (Participants) | 6 | 8 | 8 | 10 | 9 | 9 | 2 | 0 | 1 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 8 | 10 | 8 | 9 | 2 | 0 | 1 | 51
  >=65 years | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (14.3) | 46.9 (15.7) | 48.8 (12.7) | 51.6 (9.5) | 51.7 (12.4) | 50.3 (8.4) | 61.0 (1.4) |  | 52.0 (0.0) | 49.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 6 | 8 | 6 | 6 | 1 | 0 | 1 | 37
  Male | 2 | 3 | 2 | 2 | 3 | 3 | 1 | 0 | 0 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 4 | 6 | 6 | 6 | 0 | 0 | 1 | 29
  Not Hispanic or Latino | 4 | 4 | 4 | 4 | 3 | 3 | 2 | 0 | 0 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 8 | 10 | 9 | 9 | 2 |  | 1 | 53

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Insulin sensitivity in skeletal muscle (M value) as measured by hyperinsulinemic euglycemic clamp study. The clamp study tests the ability of peripheral tissues such as skeletal muscle to uptake glucose in response to a constant insulin stimulus, which give a measure of sensitivity to insulin action. 60 mU/m2*min insulin was infused into subjects for 180 minutes with concomitant adjustment of glucose infusion rate using D20 glucose to maintain a clamped plasma glucose concentration of 100 mg/dL. When the glucose infusion rate equals the rate of glucose uptake and the targeted glucose concentration is achieved, the clamp is at steady-state equilibrium. Steady-state glucose infusion rate at 150min-180mins was used as the measure to calculate the M value.
Time Frame: Change from baseline insulin sensitivity at 28 days of the intervention.
Population: Enrollment and completion for Type 2 diabetes mellitus group was low due to exclusionary criteria that prevented most diabetes medications from being used while in the study. Lean with NGT and Obese with NGT groups completed 6 control, 8 sevelamer, 8 synbiotic subjects for Lean group and 10 control, 9 sevelamer and 9 synbiotic for Obese group.
Measure: Mean (Standard Deviation); unit: M Value (mg/kg/min)
Arm/Group | Lean With NGT-Placebo | Lean With NGT-Sevelamer | Lean With NGT-Synbiotic | Obese With NGT-Placebo | Obese With NGT-Sevelamer | Obese With NGT-Synbiotic | Type 2 Diabetes-Placebo | Type 2 Diabetes-Sevelamer | Type 2 Diabetes-Synbiotic
Number analyzed (Participants) | 6 | 8 | 8 | 10 | 9 | 9 | 2 | 0 | 1
M Value (mg/kg/min) | 10.16 (3.78) | 8.45 (2.25) | 9.47 (2.59) | 5.96 (2.24) | 8.14 (2.138) | 5.45 (1.88) | 3.81 (.386) |  | 1.42
Statistical Analysis 1: Comparison: Obese With NGT-Placebo vs Obese With NGT-Sevelamer; Null hypothesis is that Sevelamer treated Obese subjects with normal glucose tolerance will show no post-treatment change in insulin sensitivity compared to placebo treated subjects; Test type: Superiority; p < 0.025, Generalized Estimating Equation — p-value not adjusted for multiple comparison, a priori threshold for significance set at p<0.025 for multiple comparisons
Statistical Analysis 2: Comparison: Obese With NGT-Placebo vs Obese With NGT-Synbiotic; Null hypothesis is that Synbiotic treated Obese subjects with normal glucose tolerance will show no post-treatment change in insulin sensitivity compared to placebo treated subjects; Test type: Superiority; p > 0.05, Generalized Estimating Equation — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Plasma Endotoxin Level and Its Panel.
Description: Plasma Lipopolysaccharide (LPS) after intervention period
Time Frame: Change from baseline plasma endotoxin level and its panel during 28 days.
Population: Poor recruitment for type 2 diabetic group means few subjects analyzed.
Measure: Mean (Standard Deviation); unit: Endotoxin units/mL
Arm/Group | Lean With NGT-Placebo | Lean With NGT-Sevelamer | Lean With NGT-Synbiotic | Obese With NGT-Placebo | Obese With NGT-Sevelamer | Obese With NGT-Synbiotic | Type 2 Diabetes-Placebo | Type 2 Diabetes-Sevelamer | Type 2 Diabetes-Synbiotic
Number analyzed (Participants) | 6 | 8 | 8 | 10 | 8 | 9 | 1 | 0 | 1
Endotoxin units/mL | 0.4452 (0.1987) | 0.5634 (0.1713) | 0.6925 (0.5907) | 0.6230 (0.1976) | 0.8012 (0.4187) | 0.7195 (0.2905) | 0.2961 |  | 0.4062
Statistical Analysis 1: Comparison: Obese With NGT-Placebo vs Obese With NGT-Sevelamer; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p > 0.05, Generalized Estimating Equation — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Obese With NGT-Placebo vs Obese With NGT-Synbiotic; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.05, Generalized Estimating Equation — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Gut Permeability
Description: urine lactulose: mannitol ratio.
Time Frame: Change from baseline gut permeability at 24 days of the intervention.
Population: One obese sevelamer subject was not able to complete their baseline Lactulose: Mannitol ratio assay, thus cannot evaluate pre-post effect from their study.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lean With NGT-Placebo | Lean With NGT-Sevelamer | Lean With NGT-Synbiotic | Obese With NGT-Placebo | Obese With NGT-Sevelamer | Obese With NGT-Synbiotic | Type 2 Diabetes-Placebo | Type 2 Diabetes-Sevelamer | Type 2 Diabetes-Synbiotic
Number analyzed (Participants) | 6 | 8 | 8 | 10 | 8 | 9 | 2 | 0 | 1
ratio | 0.02262 (0.006856) | 0.02164 (0.008943) | 0.02349 (0.008680) | 0.02055 (0.01018) | 0.01635 (0.006882) | 0.01952 (0.004869) | 0.02662 (0.004186) |  | 0.01979
Statistical Analysis 1: Comparison: Obese With NGT-Placebo vs Obese With NGT-Sevelamer; Null hypothesis is that Sevelamer treated Obese subjects with normal glucose tolerance will show no post-treatment change in Lactulose:Mannitol ratio compared to placebo treated subjects; Test type: Superiority; p > 0.05, Generalized Estimating Equation — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Obese With NGT-Placebo vs Obese With NGT-Synbiotic; Null hypothesis is that Synbiotic treated Obese subjects with normal glucose tolerance will show no post-treatment change in Lactulose:Mannitol ratio compared to placebo treated subjects; Test type: Superiority; p > 0.05, Generalized Estimating Equation — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Study participants were enrolled in the study for approximately 2-3 months.
Description: Adverse Event data was collected over the course of the subject's participation in the study, often at followup visits as part of biopsy site checks.
Arm/Group | Lean With NGT-Placebo | Lean With NGT-Sevelamer | Lean With NGT-Synbiotic | Obese With NGT-Placebo | Obese With NGT-Sevelamer | Obese With NGT-Synbiotic | Type 2 Diabetes-Placebo | Type 2 Diabetes-Sevelamer | Type 2 Diabetes-Synbiotic
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/8 | 0/10 | 0/9 | 0/9 | 0/2 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/8 | 0/10 | 0/9 | 0/9 | 0/2 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 4/6 | 3/8 | 4/8 | 6/10 | 3/9 | 4/9 | 1/2 | 0/0 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lean With NGT-Placebo (N=6) | Lean With NGT-Sevelamer (N=8) | Lean With NGT-Synbiotic (N=8) | Obese With NGT-Placebo (N=10) | Obese With NGT-Sevelamer (N=9) | Obese With NGT-Synbiotic (N=9) | Type 2 Diabetes-Placebo (N=2) | Type 2 Diabetes-Sevelamer (N=0) | Type 2 Diabetes-Synbiotic (N=1)
Biopsy Site Pain/soreness (Surgical and medical procedures) | 1 (1) | 1 (2) | 3 (3) | 3 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) — Biopsies of the vastus lateralis are obtained under local anesthesia at visit 4 and 6, before and after insulin clamp. All events expected given procedure protocol.
Fibromyalgia Exacerbation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermittent edema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Bloating/Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache/Lightheadedness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Yeast Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT02127125/Prot_SAP_000.pdf